CLINICAL TRIAL: NCT04805580
Title: Ultrasound Guided Qudratus Lumborum Block Versus Unilateral Intrathecal Block for Patient Undergoing Inguinal Hernia Repair
Brief Title: Qudratus Lumborum Block Versus Unilateral Intrathecal Block for Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hala mohamed Rashad mohamed, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Qudratus lumborum block
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Inguinal Hernia,Quadratus Lumborum Block , Unilateral Intrathecal Block
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: 2 groups (25 in each group) group intrathecal block group quadratus lumborum block
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intrathecal block (Active Comparator): patients (25) will receive unilateral intrathecal block using 1.5 ml of hyperbaric bupivacaine
  Interventions: Procedure: unilateral intrathecal block
- Quadratus lumborum block (Active Comparator): patients (25) will receive quadratus lumborum block by an anterior approach using 30 ml of bupivacaine 0.25%
  Interventions: Procedure: unilateral intrathecal block

INTERVENTIONS:
Procedure: unilateral intrathecal block — Quadratus lunborum block
  Other Names: unilateral spinal anaesthesia

SUMMARY:
compare between Quadratus lumborum block and unilateral intrathecal block for patients undergoing inguinal hernia repair regarding the quality of anesthesia and hemodynamic stability of patients.

DETAILED DESCRIPTION:
comparison between unilateral intrathecal block anesthesia (unilateral SA) and Quadratus lumborum block for inguinal hernia repair unilateral intrathecal block is widely used nowadays for unilateral inguinal hernia repair, providing intense sensory and motor blockade. Limiting the block to the operative site by using small doses of hyperbaric solutions injected slowly through a directional needle and maintaining a lateral decubitus position for a certain duration has been proposed, to produce high quality, long-duration analgesia, with minimal hemodynamic adverse events.

Previous case report studies stated that we can use Quadratus Lumborum Block as the sole anesthetic technique for open hernia repair.

ELIGIBILITY:
Inclusion Criteria:

- physical status ASA: I-II BMI >18kg/m2<30kg/m2 written informed consent from the patient scheduled for open unilateral inguinal hernia repair

Exclusion Criteria:

* uncooperative patient
* Allergy to local anesthetic drugs
* patients on chronic alcohol, opioid, tranquilizer or sedative use
* Pregnant females.
* Psychological, mental disorders, or depression.
* Patients receiving anticoagulants therapy or suspected coagulopathy.
* Patients with infection or previous surgery at sit of anesthetic procedures.
* Patients with significant cardiovascular, respiratory, renal, hepatic, or metabolic disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
To assess safety of quadratus lumborum block vs unilateral intrathecal block for inguinal hernia repair: complications of the block | 2 hours
  complications of the block in each group like inadequate blockade detected by increased dose of sedation required in this group ,hemodynamic instability related to the block detected by frequent monitoring of the blood pressure and heart rate

SECONDARY OUTCOMES:
To compare the onset and duration of sensory block between both blocks | 12 hours
  the onset of pin brick discrimination and time of first request of analgesics after block performance in each group
To compare the time to ambulation | 24 hours
  the time till the patient succeed in ambulation

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 1 year

REFERENCES:
- [Background] Favaro ML, Gabor S, Souza DBF, Araujo AA, Milani ALC, Ribeiro Junior MAF. Quadratus Lumborum Block As A Single Anesthetic Method For Laparoscopic Totally Extraperitoneal (Tep) Inguinal Hernia Repair: A Randomized Clinical Trial. Sci Rep. 2020 May 22;10(1):8526. doi: 10.1038/s41598-020-65604-x. PMID 32444629
- [Background] La Colla L, La Colla MDL, Schroeder R, Schroeder RMD. Quadratus Lumborum Block as Sole, Homeostatic-Preserving Anesthetic for a Patient with Multiple System Atrophy Undergoing Open Inguinal Hernia Repair: A Case Report. Case Rep Anesthesiol. 2018 Jun 28;2018:7161860. doi: 10.1155/2018/7161860. eCollection 2018. PMID 30050698
- [Background] Isil CT, Cinar AS, Oba S, Isil RG. Comparison of Spinal Anaesthesia and Paravertebral Block in Unilateral Inguinal Hernia Repair. Turk J Anaesthesiol Reanim. 2014 Oct;42(5):257-63. doi: 10.5152/TJAR.2014.75508. Epub 2014 Jul 9. PMID 27366432